CLINICAL TRIAL: NCT01370200
Title: Regional Citrate Anticoagulation in Plasma Exchange Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Manja Antonic, MD, University Medical Centre Ljubljana
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 111/09/09
Record Dates: First submitted 2011-06-02; First posted 2011-06-09 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-05

CONDITIONS: Focal Segmental Glomerulosclerosis; Guillain-Barre Syndrome
Keywords: citrate; anticoagulation; plasma exchange; efficacy
MeSH Terms: conditions — Glomerulosclerosis, Focal Segmental; Guillain-Barre Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 4% citrate (Active Comparator): 4% trisodium citrate, starting infusion rate 180 ml/h Interventions according to postfilter ionized calcium, change in 10 ml/h step
  Interventions: Procedure: plasma exchange treatment
- 15% citrate (Active Comparator): 15% trisodium citrate, starting infusion rate 50 ml/h Interventions according to postfilter ionized calcium, change in 10 ml/h step
  Interventions: Procedure: plasma exchange treatment

INTERVENTIONS:
Procedure: plasma exchange treatment — the therapeutic plasma exchange is the procedure of removing the plasma of the patient including pathological macromolecules and replacing it with the replacement fluid

SUMMARY:
The investigators want to compare the efficacy of plasma exchange treatment with using two different citrates ( 4% and 15% ) as anticoagulants in plasma exchange treatment.

The efficacy of plasma exchange treatment is better with using 15% trisodium citrate as anticoagulant during the plasma exchange procedure.

DETAILED DESCRIPTION:
To compare the elimination rate of immunoglobulins in plasma exchange treatment by using two differently concentrated citrates for anticoagulation during plasma exchange procedure. At the same time we want to compare acid-base , electrolyte status and anticoagulation protocol in two citrate groups.

ELIGIBILITY:
Inclusion Criteria:

* patients who need plasma exchange treatment
* human albumins as a replacement fluid

Exclusion Criteria:

* anemia Hb less than 90

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2011-04; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
The efficacy of plasma exchange, measuring immunoglobulins type G before and after the procedure, using 4% and 15% citrate as anticoagulants | the whole trial, approximately 3 years

SECONDARY OUTCOMES:
The percentage of patients in whom there is a 50% reduction of immunoglobulins after plasma exchange using 4% and 15% citrate as anticoagulants | the whole trial, approximately 3 years
Using 15% citrate as an anticoagulant during plasma exchange treatment is as safe as using 4% citrate as anticoagulant during plasma exchange treatment. | the whole trial, approximately 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Manja Antonič, MD, Principal Investigator — Center for acute and complicated dialysis, UMCLjubljana
Locations (1):
- Center for acute and complicated dialysis, Clinical department of nephrology, UMC Ljubljana, Ljubljana, Slovenia

REFERENCES:
- [Background] Antonic M, Gubensek J, Buturovic-Ponikvar J, Ponikvar R. Comparison of citrate anticoagulation during plasma exchange with different replacement solutions. Ther Apher Dial. 2009 Aug;13(4):322-6. doi: 10.1111/j.1744-9987.2009.00733.x. PMID 19695068